CLINICAL TRIAL: NCT04679597
Title: Total Neoadjuvant Therapy Versus Standard Therapy of Locally Advanced Rectal Cancer With High Risk Factors for Failure
Status: Completed | Type: Observational
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: ERID-KSOPKR-0009/2019
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- total neoadjuvant therapy: Total neoadjuvant therapy consisted of 12 weeks of induction chemotherapy with CAPOX or FOLFOX, chemoradiotherapy with capecitabine and six to eight weeks of consolidation chemotherapy with CAPOX or FOLFOX prior to surgery.
  Interventions: Drug: Capecitabine
- standard therapy: Standard therapy (neoadjuvant chemoradiotherapy, surgery, adjuvant chemotherapy)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — comparison of two treatments
  Other Names: oxaliplatin

SUMMARY:
In a retrospective study, the investigators will compare patients with locally advanced rectal cancer with high risk factors for failure who were treated with standard therapy or with total neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven locally advanced rectal cancer and
* the presence of one of the factors: T4, N2, positive mesorectal fascia, presence of extramural vascular invasion or presence of lateral lymph node.

Exclusion Criteria:

* distant metastases,
* concomitant malignancy,
* inflammatory bowel disease, or
* malabsorption syndrome.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adult patients with newly diagnosed LARC with high risk factors for failure who were treated with TNT or standard therapy at the Institute of Oncology, Ljubljana, from 2016 to 2019
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
pathological complete response | during surgery
  pathological complete response is defined as the absence of tumor cells in the surgical resection

SECONDARY OUTCOMES:
Neoadjuvant rectal cancer score | during treatment, assessed up to 10 days
  Neoadjuvant rectal cancer score: The NAR score was calculated using the equation [5 pN - 3(cT - pT) + 12]^2 / 9.61 and further classified as low (< 8), intermediate (8-16), or high (< 16).

OTHER OUTCOMES:
number of participants who completed treatment | during treatment, assessed up to 10 days
  Compliance - number of participants who completed treatment protocol
number of participants with acute side effects | during treatment, assessed up to 10 days
  Acute toxcity - number of participants with side effects during different treatment modality